CLINICAL TRIAL: NCT05506020
Title: Retrospective Study on the Application of ICG Fluorescence Cholangiography in Laparoscopic Living Donor Left Lateral Sectionectomy
Brief Title: Application of ICG Fluorescence Cholangiography in Laparoscopic Living Donor Left Lateral Sectionectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lunxiu Qin, Director of the department of general surgery, Huashan Hospital, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Huashan009
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Living Donor Liver Transplantation
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICG group (Experimental): indocyanine green (ICG) fluorescence cholangiography
  Interventions: Procedure: indocyanine green (ICG) fluorescence cholangiography
- non ICG group (No Intervention): no intervention

INTERVENTIONS:
Procedure: indocyanine green (ICG) fluorescence cholangiography — indocyanine green (ICG) fluorescence cholangiography during operation
  Arms: ICG group

SUMMARY:
The purpose of this study was to assess the effects of indocyanine green (ICG) fluorescence cholangiography during laparoscopic left lateral sectionectomy (LLLS) on the occurrence of biliary complications in both donors and recipients in living donor liver transplantation (LDLT) and to explore the optimal dose and injection time of ICG.

DETAILED DESCRIPTION:
This was a retrospective cohort study. The purpose of this study was to assess the effects of indocyanine green (ICG) fluorescence cholangiography during LLLS on the occurrence of biliary complications in both donors and recipients. The optimal dose and injection time of ICG were also investigated. From October 2016 to May 2022, the clinical data of 85 donors who underwent LLLS and relevant recipients in the Department of General Surgery of Huashan Hospital were retrospectively analyzed. According to whether ICG fluorescence cholangiography was used, they were divided into a non-ICG group (n=46) and an ICG group (n=39). Biliary complications were observed and the optimal dose and injection time of ICG were explored.

ELIGIBILITY:
Inclusion Criteria:

1. From October 2016 to May 2022, donors and their corresponding recipients underwent laparoscopic donor liver acquisition surgery in the general surgery department of Huashan Hospital.
2. Donor age ≥ 18 years old, regardless of gender; The receptor is the corresponding receptor of the donor, and the age and sex of the receptor are unlimited.
3. The medical history is complete, which can meet the requirements of this study.
4. Volunteer to participate in this study.

Exclusion Criteria:

1. The medical history is incomplete, which cannot meet the requirements of this study.
2. The donor or recipient expressly refused to participate in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2022-07 (Actual)

PRIMARY OUTCOMES:
Biliary complications | two months after operation
  bile leakage and biliary stenosis

CONTACTS AND LOCATIONS:
Overall Officials: Lunxiu Qin, Principal Investigator — Department of general surgery, Huashan Hospital

IPD SHARING:
Plan to Share IPD: No